CLINICAL TRIAL: NCT00707681
Title: A Phase II Randomized, Controlled Study to Evaluate the Quality of Life, Survival and Therapeutic Benefits of MS-20 in Patient With Advanced Hepatocellular Carcinoma
Brief Title: Evaluation of Quality of Life and Survival With MS-20 in Patient With Advanced Hepatocellular Carcinoma (FDA IND 74572)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Microbio Co Ltd (Industry)
Responsible Party: Mr. David Yeh, Director, MicroBio Co., Ltd.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MCRA06001A
Record Dates: First submitted 2008-06-30; First posted 2008-07-01 (Estimated); Last update posted 2010-02-26 (Estimated); Status verified 2010-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: microbio, MS-20, Hepatoma, Advanced Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (Active Comparator): MS-20
  Interventions: Drug: MS-20
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MS-20 — 4 ml/vial
  Arms: I
Drug: Placebo — 4ml/vial
  Arms: 2

SUMMARY:
To evaluate Quality of Life (QoL) score of MS-20 versus placebo in advanced HCC patients using European Organization for Research and Treatment of Cancer (EORTC) QLQ C-30 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

Subjects may be included in the study only if they meet all of the following criteria:

1. Subject aged ≧ 20;
2. Histologically documented, unresectable advanced HCC. For patients with difficulty in obtaining histological diagnosis, a "clinical diagnosis" of HCC is acceptable if all the following criteria are met:

   * Chronic hepatitis B or C with evidence of liver cirrhosis;
   * Presence of hepatic tumor(s) with image findings (sonography, CT scan) compatible with HCC and no evidence of gastrointestinal tumors;
   * Elevated serum α-fetoprotein level ≧ 400 ng/ml;
3. Cancer of the Liver Italian Program (CLIP) score of 3-4;
4. Liver transaminase ≦ 5 times upper normal limits (UNL);
5. Patient fulfilling any of the follow conditions:

   * Refuse to receive aggressive cancer therapy after explained to the subjects the benefits and risks;
   * Progressive malignant disease after previous radiotherapy, percutaneous ethanol injection, radiofrequency ablation, transarterial embolization, transarterial chemoembolization, systemic chemotherapy, immunotherapy, or any experimental therapy, or unable to tolerate such therapy;
   * No treatment of high priority is available;
6. ECOG performance status of 0 - 2;
7. Patients are willing and able to comply with study procedures and sign informed consent.

Exclusion Criteria

Subjects will be excluded from the study for any of the following reasons:

1. Patient with history of HCC rupture;
2. Medical condition requiring anticoagulant or anti-platelet drugs;
3. Patients with brain metastases;
4. Patient unable to receive oral medication;
5. Patients with significant renal function impairment (creatinine>1.5mg/dl), severe cardiac disease, e.g. angina pectoris, myocardial infarction, cardiac arrhythmia, congestive heart failure (New York Heart Association Functional Classification III and IV) or physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that might render the subject at high risk from treatment;
6. Female subjects of childbearing potential who:

   * are lactating; or
   * have positive pregnancy test (urine) at V2;
7. Active infection or on antiretroviral therapy for HIV disease;
8. Patient with known hypersensitivity to any component of the study medication (soy bean or soy product).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate Quality of Life (QoL) score of MS-20 versus placebo in advanced HCC patients | 24 weeks

SECONDARY OUTCOMES:
Overall survival, Overall survival rate, Change from baseline of the highest weight observed, Change from baseline of body weight | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Yuan Peng, MD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan